CLINICAL TRIAL: NCT02663518
Title: A Phase 1a/1b Dose Escalation and Expansion Trial of TTI-621, a Novel Biologic Targeting CD47, in Subjects With Relapsed or Refractory Hematologic Malignancies and Selected Solid Tumors
Brief Title: A Trial of PF-07901800 (TTI-621) for Patients With Hematologic Malignancies and Selected Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer decided terminating study for administrative reasons on 22Mar2022 (stopping enrollment as of 15Apr2022). The decision wasn't due to safety concerns or requests from regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTI-621-01; C4961001 (Other: Alias Study Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancies; Solid Tumor
Keywords: PF-07901800; ABCL; Aggressive B-cell lymphoma; CLL; Chronic lymphocytic leukemia; CTCL; Cutaneous T-Cell Lymphoma; HL; Hodgkin lymphoma; IBCL; Indolent B-cell lymphoma; MDS; Myelodysplastic syndromes; MPN; Myeloproliferative neoplasms; MM; Multiple Myeloma; PTCL; Peripheral T-cell lymphomas; SCLC; Small Cell Lung Cancer; T-cell lymphoma; Rituximab; Nivolumab; TTI-621; Solid Tumor; Hematologic Malignancies; Lymphoma; CD47; SIRPα-IgG1 Fc
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Hodgkin Disease; Myelodysplastic Syndromes; Myeloproliferative Disorders; Multiple Myeloma; Lymphoma, T-Cell, Peripheral; Small Cell Lung Carcinoma; Lymphoma, T-Cell; Lymphoma | interventions — TTI-621; Rituximab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase 1a/1b trial of PF-07901800 (TTI-621) for relapsed or refractory hematologic malignancies and selected solid tumors were conducted in 4 parts. In the dose escalation phase (Part 1), advanced lymphomas were enrolled in sequential dose cohorts for safety, tolerability, PK, and MTD. In the expansion phase (Part 2), subjects with various hematologic malignancies and selected solid tumors were treated at recommended dose determined in phase 1a (Part 1) for safety and efficacy. In the expansion phase (Part 3), 2 cohorts (cutaneous T-cell lymphoma and peripheral T-cell lymphoma) were evaluated for potentially further studied using Simon 2-stage design. In the phase 1b dose optimization (Part 4), further dose escalation was investigated in patients with relapsed and/or refractory CTCL following a 3+3 escalation and revised DLT criteria.
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (16):
- PF-07901800 (TTI-621) Escalation Phase - R/R Lymphoma (Experimental): The Escalation Phase will include multiple doses of PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Indolent B-Cell Lymphoma (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Aggressive B-Cell Lymphoma (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- T-Cell Lymphoma (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Hodgkin Lymphoma (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Chronic Lymphocytic Leukemia (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Multiple Myeloma (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Acute Myeloid Leukemia (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Myelodysplastic Syndrome (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Myeloproliferative Neoplasms (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Small Cell Lung Cancer (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Rituximab Combination (Experimental): Combination therapy expansion cohort with PF-07901800 (TTI-621) plus Rituximab for CD20 positive malignancies
  Interventions: Drug: PF-07901800 (TTI-621) plus Rituximab
- Nivolumab Combination (Experimental): Combination therapy expansion cohort with PF-07901800 (TTI-621) plus Nivolumab for Hodgkin Lymphoma
  Interventions: Drug: PF-07901800 (TTI-621) plus Nivolumab
- Cutaneous T-Cell Lymphoma (CTCL) (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Peripheral T-Cell Lymphoma (PTCL) (Experimental): Monotherapy expansion cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)
- Part 4: Cutaneous T-Cell Lymphoma (CTCL) (Experimental): Monotherapy expansion Part 4 (Dose Optimization) cohort with PF-07901800 (TTI-621)
  Interventions: Drug: PF-0791800 (TTI-621)

INTERVENTIONS:
Drug: PF-0791800 (TTI-621) — Monotherapy
  Other Names: TTI-621 (SIRPα-IgG1 Fc)
  Arms: Acute Myeloid Leukemia; Aggressive B-Cell Lymphoma; Chronic Lymphocytic Leukemia; Cutaneous T-Cell Lymphoma (CTCL); Hodgkin Lymphoma; Indolent B-Cell Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome; Myeloproliferative Neoplasms; PF-07901800 (TTI-621) Escalation Phase - R/R Lymphoma; Part 4: Cutaneous T-Cell Lymphoma (CTCL); Peripheral T-Cell Lymphoma (PTCL); Small Cell Lung Cancer; T-Cell Lymphoma
Drug: PF-07901800 (TTI-621) plus Rituximab — Combination therapy
  Other Names: TTI-621 plus Rituxan
  Arms: Rituximab Combination
Drug: PF-07901800 (TTI-621) plus Nivolumab — Combination therapy
  Other Names: TTI-621 plus Opdivo
  Arms: Nivolumab Combination

SUMMARY:
Multicenter, open-label, phase 1a/1b trial of PF-07901800 (TTI-621) in subjects with relapsed or refractory hematologic malignancies and selected solid tumors.

DETAILED DESCRIPTION:
This is a trial of PF-07901800 (TTI-621) in subjects with relapsed or refractory hematologic malignancies and selected solid tumors.

TTI-621 (SIRPαFc) is a soluble recombinant fusion protein created by directly linking the sequences encoding the N-terminal CD47 binding domain of human SIRPα with the Fc domain of human immunoglobulin (IgG1). TTI-621 acts by binding human CD47 and preventing it from delivering an inhibitory "do not eat" (anti phagocytic) signal to macrophages.

This trial will be conducted in 2 phases and 4 parts: Phase 1a Part 1 (escalation phase) and Phase 1b Parts 2-4 (expansion phase).

In the dose Escalation Phase (phase 1a Part 1), subjects with lymphoma will be enrolled in sequential dose cohorts to receive TTI-621 to characterize safety, tolerability, pharmacokinetics, and the maximum-tolerated dose (MTD).

In the Expansion Phase (phase 1b Parts 2-4), TTI-621 will be given to subjects with a variety of hematologic malignancies and selected solid tumors to further define safety and to characterize efficacy. In the Expansion Phase Part 2, the safety and efficacy of TTI-621 will also be assessed when it is given in combination with other anti-cancer drugs. The dose of TTI-621 to be delivered in the Expansion Phase Parts 2-3 of the study may be increased or decreased based on the subject's tolerability and on the subject's response to treatment.

In the phase 1b dose optimization of the study (Part 4), further dose escalation of TTI-621, beyond the dose determined during phase 1a dose escalation, will be pursued in patients with relapsed and/or refractory CTCL following a 3+3 escalation design and using a revised DLT criteria to further evaluate the safety and tolerability of TTI-621 at dose levels higher than the initially recommended phase 1b Parts 2-3.

Secondary objectives include further characterization of the pharmacokinetics, pharmacodynamics, and development of ADA; and to gain preliminary evidence of the anti-tumor activity of TTI-621 in subjects with a variety of hematologic malignancies and selected solid tumors. In addition, the safety of TTI-621 will be evaluated in combination with other anti-cancer agents.

Pfizer decided terminating this study for administrative reasons on 22Mar2022 (stopping enrollment as of 15Apr2022). The decision wasn't due to safety concerns or requests from regulatory authorities.

ELIGIBILITY:
MAJOR ELIGIBILITY CRITERIA:

Phase 1a Escalation

• Histologically documented, measurable, advanced lymphomas, transfusion-independence

Phase 1b Expansion (Part 2 and 3) • Advanced malignancy: IBCL, ABCL, cHL, AML, ALL, MDS, MPN, SCLC, PTCL and CTCL; measurable disease who have relapsed or are refractory following at least 2 prior systemic therapeutic attempts (1 prior systemic attempt for PTCL). For CTCL, extracorporeal photochemotherapy (ECP) considered a systemic therapy. Local radiation and topical agents are not systemic therapies.

Phase 1b dose optimization (Part 4)

• Histologically confirmed diagnosis of CTCL (both Mycosis Fungoides and Sezary Syndrome): Failed at least 2 prior systemic therapies for CTCL (Systemic therapy does not include local radiation therapy or topical agents); History of histologically documented diagnosis of CTCL stage IB to IVB

Inclusion Criteria (all subjects):

* Advanced measurable malignancy with previously progressed on, or currently progressing on standard anticancer therapy or for whom no other approved conventional therapy exists
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Adequate hematologic, hepatic, renal, and coagulation function; fresh or archived tumor tissue available for immunohistochemistry
* Recovery from prior treatments and/or surgeries; no history of hemolytic anemia or bleeding diathesis.
* AML M3 (French American British, FAB, classification) (i.e., acute promyelocytic leukemia [APL]) excluded

Exclusion Criteria:

* Known current central nervous system disease involvement or untreated brain metastases
* Allogeneic transplant within 30 days prior to the planned start of treatment or subjects with active graft-vs-host disease with the exception of Grade 1 skin involvement
* History of hemolytic anemia or bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (47):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope, Duarte, California
  - Freidenrich Center for Translational Research (CTRU), Palo Alto, California
  - Stanford Cancer Institute, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian/St.Luke's Medical Center, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center Richard M Schulze Family Foundation Outpatient Center at McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Covance Biorepository, Greenfield, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack Meridian Health John Theurer Cancer Center, Hackensack, New Jersey
  - Hackensack UMC, Hackensack, New Jersey
  - The John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYU Investigational Pharmacy, New York, New York
  - NYU Langone Health (Tisch Hospital), New York, New York
  - Memorial Sloan Kettering Cancer Center-Clinical Trails Office, New York, New York
  - Columbia Univeristy, New York, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care, New York, New York
  - Memorial Sloan Kettering Cancer Center Rockefeller Outpatient Pavillion, New York, New York
  - Columbia University Medical Center., New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University-Research Pharmacy Services, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pittsburgh Medical Center Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee
  - Sarah Cannon Research Institute (Pharmacy), Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Myriad RMB Inc, Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Cancer Prevention Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Melanoma and Skin Clinic, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Canada (4):
  - Fairmont Medical Building, Suite 810, Vancouver, B.C.
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Marks JA, Wang X, Fenu EM, Bagg A, Lai C. TP53 in AML and MDS: The new (old) kid on the block. Blood Rev. 2023 Jul;60:101055. doi: 10.1016/j.blre.2023.101055. Epub 2023 Feb 14. PMID 36841672
- [Derived] Ansell SM, Maris MB, Lesokhin AM, Chen RW, Flinn IW, Sawas A, Minden MD, Villa D, Percival MM, Advani AS, Foran JM, Horwitz SM, Mei MG, Zain J, Savage KJ, Querfeld C, Akilov OE, Johnson LDS, Catalano T, Petrova PS, Uger RA, Sievers EL, Milea A, Roberge K, Shou Y, O'Connor OA. Phase I Study of the CD47 Blocker TTI-621 in Patients with Relapsed or Refractory Hematologic Malignancies. Clin Cancer Res. 2021 Apr 15;27(8):2190-2199. doi: 10.1158/1078-0432.CCR-20-3706. Epub 2021 Jan 15. PMID 33451977
- [Derived] Johnson LDS, Banerjee S, Kruglov O, Viller NN, Horwitz SM, Lesokhin A, Zain J, Querfeld C, Chen R, Okada C, Sawas A, O'Connor OA, Sievers EL, Shou Y, Uger RA, Wong M, Akilov OE. Targeting CD47 in Sezary syndrome with SIRPalphaFc. Blood Adv. 2019 Apr 9;3(7):1145-1153. doi: 10.1182/bloodadvances.2018030577. PMID 30962222
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TTI-621-01

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 249 participants were enrolled in the study.
Groups:
- Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.05 milligram per kilogram (mg/kg) infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.1 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.2 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.3 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 2: Participants with a broader variety of hematologic malignancies and selected solid tumors, received a 0.2 mg/kg/week TTI-621 infusion until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination: Participants with Classical Hodgkin's Lymphoma (cHL) received 0.1 mg/kg/week TTI-621 infusion along with 3 mg/kg nivolumab given every 2 weeks or a fixed dose per current FDA approved package insert for cHL. If required dose of TTI-621 could be increased up to 0.5 mg/kg/week. Participants received TTI-621 monotherapy upon completion of combination partner regimen/unacceptable toxicity to the combination regimen.
- Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination: Participants with CD20-positive malignancies received 0.1 mg/kg/week TTI-621 infusion along with 375 milligram per meter square (mg/m^2) rituximab given weekly (1 cycle) for up to 8 cycles according to the institutional standard of care. Participants received TTI-621 monotherapy upon completion of combination partner regimen/unacceptable toxicity to the combination regimen.
- Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 3: Participants with cutaneous T-cell lymphoma (CTCL) and peripheral T-cell lymphoma (PTCL), received a 0.2 mg/kg/week TTI-621 infusion. Initial 2 weeks of 0.2 mg/kg treatment followed by intraparticipant dose intensification at an increment of 0.1 mg/kg per week up to 0.5 mg/kg within 5-8 weeks until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 0.5 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 0.7 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 1.0 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 1.4 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 2.0 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg: Participants with relapsed or refractory CTCL received a 2.0 mg/kg TTI-621 infusion once every 2 weeks until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
Period: Part 1: Phase 1a Escalation
Arm/Group | Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 2 | Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 3 | Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Started | 3 (Part 1 participants.) | 3 (Part 1 participants.) | 7 (Part 1 participants.) | 5 (Part 1 participants.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 and 3: Phase 1b Expansion
Arm/Group | Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 2 | Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 3 | Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Started | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 107 (Part 2 participants.) | 11 (Part 2 participants.) | 40 (Part 2 participants.) | 42 (Part 3 participants.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.) | 0 (No participants for part 2 and 3.)
Completed | 0 | 0 | 0 | 0 | 29 | 10 | 6 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 78 | 1 | 34 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 50 | 0 | 25 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 0 | 0 | 0 | 0 | 16 | 1 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4: Phase 1b Dose Optimization
Arm/Group | Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 2 | Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Ontorpacept (PF-07901800/TTI-621) Monotherapy for Part 3 | Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Started | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 0 (No participants for part 4.) | 3 (Part 4 participants.) | 3 (Part 4 participants.) | 6 (Part 4 participants.) | 3 (Part 4 participants.) | 12 (Part 4 participants.) | 4 (Part 4 participants.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 8 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Informed Consent Withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all the participants who received at least one dose of study treatment.
Groups:
- Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.05 milligram per kilogram (mg/kg) infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.1 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.2 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.3 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy: Participants with a broader variety of hematologic malignancies and selected solid tumors, received a 0.2 mg/kg/week TTI-621 infusion until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination: Participants with cHL received 0.1 mg/kg/week TTI-621 infusion along with 3 mg/kg nivolumab given every 2 weeks or a fixed dose per current FDA approved package insert for cHL.If required dose of TTI-621 could be increased up to 0.5 mg/kg/week. Participants received TTI-621 monotherapy upon completion of combination partner regimen/unacceptable toxicity to the combination regimen.
- Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination: Participants with CD20-positive malignancies received 0.1 mg/kg/week TTI-621 infusion along with 375 mg/m^2 rituximab given weekly (1 cycle) for up to 8 cycles according to the institutional standard of care. Participants received TTI-621 monotherapy upon completion of combination partner regimen/unacceptable toxicity to the combination regimen.
- Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy: Participants with CTCL and PTCL, received a 0.2 mg/kg/week TTI-621 infusion. Initial 2 weeks of 0.2 mg/kg treatment followed by intraparticipant dose intensification at an increment of 0.1 mg/kg per week up to 0.5 mg/kg within 5-8 weeks until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 0.5 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 0.7 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 1.0 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 1.4 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 2.0 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg: Participants with relapsed or refractory CTCL received a 2.0 mg/kg TTI-621 infusion once every 2 weeks until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Total: Total of all reporting groups
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 7 | 5 | 107 | 11 | 40 | 42 | 3 | 3 | 6 | 3 | 12 | 4 | 249
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 2 | 3 | 6 | 2 | 52 | 11 | 19 | 20 | 2 | 2 | 3 | 0 | 7 | 1 | 130
  65 - < 75 Years | 1 | 0 | 1 | 3 | 36 | 0 | 17 | 11 | 0 | 1 | 0 | 2 | 1 | 1 | 74
  75 - < 85 Years | 0 | 0 | 0 | 0 | 19 | 0 | 4 | 10 | 1 | 0 | 3 | 1 | 4 | 1 | 43
  >= 85 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 46 | 5 | 10 | 18 | 1 | 1 | 4 | 0 | 2 | 1 | 96
  Male | 2 | 2 | 4 | 2 | 61 | 6 | 30 | 24 | 2 | 2 | 2 | 3 | 10 | 3 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 0 | 8 | 2 | 4 | 5 | 0 | 1 | 0 | 0 | 1 | 0 | 26
  Not Hispanic or Latino | 3 | 3 | 2 | 5 | 94 | 9 | 34 | 32 | 3 | 2 | 5 | 3 | 11 | 3 | 209
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 5 | 0 | 0 | 1 | 0 | 0 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 6 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 12 | 1 | 1 | 7 | 1 | 1 | 0 | 0 | 2 | 1 | 28
  White | 3 | 0 | 5 | 5 | 85 | 10 | 31 | 30 | 2 | 1 | 5 | 3 | 9 | 2 | 191
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 3 | 0 | 3 | 4 | 0 | 1 | 1 | 0 | 1 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in administered medicinal product, event need not necessarily have a causal relationship with product treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. Treatment emergent AEs were events emerged during treatment period and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part 1: Day 1 of dosing up to 30 days of safety follow-up visit after the last dose (maximum treatment exposure for Part 1 was 414 days)
Population: Safety population included all the participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.05 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 3 | 3 | 7 | 5
Participants
  TEAEs | 3 | 3 | 7 | 5
  TESAEs | 1 | 0 | 1 | 2

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the protocol specified TEAEs that occurred during the 21-day. DLT treatment/observation period (including the pre-dose tests on Day 22/Week 4 Day 1) and that were considered at least possibly related to study treatment by the investigator. Protocol specified DLT TEAE criteria: Grade 4 thrombocytopenia; Grade 3 thrombocytopenia with bleeding (with the exception of brief, easily-controlled epistaxis, mild gum bleeding or normal menses) or with any requirement for platelet transfusions; Grade 4 anemia, unexplained by underlying disease; Grade 4 neutropenia lasting more than 5 days; Febrile neutropenia of any duration ( Absolute Neutrophil Count (ANC) less than (<) 1.0 * 10^9/L. fever greater than (>) 38.5° Degree Celsius (C); Grade 3 or higher non-hematologic toxicity except for alopecia and nausea controlled by medical management; Grade 3 or 4 hemorrhage.
Time Frame: Part 1: Day 1 of dosing up to Pre-dose on Day 22
Population: The DLT-evaluable set included participants who had received all 3 doses within the DLT evaluation period, or participants who experienced an AE, meeting DLT criteria during that time. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 5
Participants | 0 | 0 | 1 | 2

3. Primary Outcome: Part 2 and 3: Number of Participants With TEAEs and TESAEs
Description: An AE was any untoward medical occurrence in administered medicinal product, event need not necessarily have a causal relationship with product treatment or usage. A SAE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. Treatment emergent AEs were events emerged during treatment period and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 of dosing up to 30 days of safety follow-up visit after the last dose (maximum treatment exposure for Part 2 was 1793 days and for Part 3 was 938 days)
Population: Analysis population included all the participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination: Participants with cHL received 0.1 mg/kg/week TTI-621 infusion along with 3 mg/kg nivolumab given every 2 weeks or a fixed dose per current FDA approved package insert for cHL. If required dose of TTI-621 could be increased up to 0.5 mg/kg/week. Participants received TTI-621 monotherapy upon completion of combination partner regimen/unacceptable toxicity to the combination regimen.
Arm/Group | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination
Number analyzed (Participants) | 107 | 42 | 11 | 40
Participants
  TEAEs | 103 | 40 | 11 | 37
  TESAEs | 43 | 15 | 2 | 13

4. Primary Outcome: Part 4: Number of Participants With TEAEs and TESAEs
Description: An AE was any untoward medical occurrence in administered medicinal product, event need not necessarily have a causal relationship with product treatment or usage. A SAE event was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. Treatment emergent AEs were events emerged during treatment period and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part 4: Day 1 of dosing up to 1 year of safety follow-up visit after the last dose (maximum treatment exposure for Part 4 was 667 days)
Population: Analysis population included all the participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 4: TTI-621 2 mg/kg: Participants with relapsed or refractory CTCL received TTI-621 2 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: TTI-621 2 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 4
Participants
  TEAEs | 3 | 3 | 6 | 3 | 12 | 4
  TESAEs | 1 | 1 | 2 | 0 | 3 | 3

5. Primary Outcome: Part 4: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the protocol specified TEAEs that occurred during the 21-day. DLT treatment/observation period (including the pre-dose tests on Day 22/Week 4 Day 1) and that were considered at least possibly related to study treatment by the investigator. Protocol specified DLT TEAE criteria: Grade 4 thrombocytopenia; Grade 3 thrombocytopenia with bleeding (with the exception of brief, easily-controlled epistaxis, mild gum bleeding or normal menses) or with any requirement for platelet transfusions; Grade 4 anemia, unexplained by underlying disease; Grade 4 neutropenia lasting more than 5 days; Febrile neutropenia of any duration (ANC < 1.0 x 109/L, fever > 38.5°C); Grade 3 or higher non-hematologic toxicity except for alopecia and nausea controlled by medical management; Grade 3 or 4 hemorrhage.
Time Frame: Part 4: Day 1 of dosing up to Pre-dose on Day 22
Population: The DLT-evaluable set included participants who had received all 3 doses within the DLT evaluation period, OR participants who experienced an AE, meeting DLT criteria during that time. As 2.0mg/kg Q2W cohort was not a part of escalation for dose optimization, and not relevant to DLT assessment hence this outcome measure was not analyzed for Q2W arm. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: TTI-621 2 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 7 | 0
Participants | 0 | 0 | 1 | 0 | 2 |

6. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of TTI-621
Time Frame: Part 1: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: Pharmacokinetic (PK)-evaluable set included treated participants with adequate blood sampling to estimate at least one pharmacokinetic PK parameter.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 3 | 3 | 7 | 5
Nanogram per milliliter | 136.594 (64.248) | 366.636 (67.433) | 823.137 (153.681) | 1579.799 (518.546)

7. Secondary Outcome: Part 1: Area Under the Plasma Concentration Time Curve From Time Zero to 168 (AUC[0-168]) of TTI-621
Time Frame: Part 1: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: PK evaluable set included treated participants with adequate blood sampling to estimate at least one pharmacokinetic PK parameter. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram*hour/milliliter
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 1 | 2 | 5 | 4
Nanogram*hour/milliliter | 1200.722 | 6178.488 (844.463) | 18873.939 (6213.503) | 36782.700 (8700.626)

8. Secondary Outcome: Part 1: Percentage of CD47 Receptor Occupancy on Peripheral Blood CD3+ Cells
Description: CD47 is a cell-surface protein expressed on multiple normal cell types and often at high levels on many malignant tumour cells .
Time Frame: Part 1: Week 1 end of infusion (EOI)
Population: This outcome measure was not analyzed since CD47 data for Part 1 was not collected as the assay was not set up when enrolling the Part 1 participants. Hence, no participants evaluable for this outcome measure.
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Part 1: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb)
Description: A participant was ADA (or NAb) positive if: (1) baseline titer was missing or negative and participants had >1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a > [4-fold dilution increase] in titer from baseline in >1 post-treatment sample (treatment-boosted).
Time Frame: Part 1: From pre-infusion on day 1 up to end of study treatment (maximum treatment exposure for Part 1 was 414 days)
Population: Immunogenicity analysis population included all treated participants with at least one ADA sample (pre-dose or post-treatment) analyzed. Here, "Number of Participants Analyzed" signifies number of participants who were ADA or NAb evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg
Number analyzed (Participants) | 3 | 3 | 7 | 4
Participants
  ADA Positive: Overall Incidence | 1 | 0 | 1 | 0
  NAb Positive: Overall Incidence | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 2 and 3 Combined: Maximum Plasma Concentration (Cmax) of TTI-621
Description: Results for this outcome measure was reported for Part 2 and Part 3 combined.
Time Frame: Part 2 and 3: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: PK evaluable set included treated participants with adequate blood sampling to estimate at least one PK parameter. Here, "Number of participants analyzed" signifies number of evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Groups:
- Part 2 and 3 Combined: 0.1 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.1 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2 and 3 Combined: 0.2 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.2 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2 and 3 Combined: 0.3 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.3 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2 and 3 Combined: 0.4 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.4 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2 and 3 Combined: 0.5 mg/kg: Participants with advanced relapsed or refractory CTCL received TTI-621 0.5 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
Arm/Group | Part 2 and 3 Combined: 0.1 mg/kg | Part 2 and 3 Combined: 0.2 mg/kg | Part 2 and 3 Combined: 0.3 mg/kg | Part 2 and 3 Combined: 0.4 mg/kg | Part 2 and 3 Combined: 0.5 mg/kg
Number analyzed (Participants) | 50 | 147 | 0 | 1 | 0
Nanogram per milliliter | 341 (160) | 1020 (1270) |  | 673 |

11. Secondary Outcome: Part 2 and 3 Combined: Area Under the Plasma Concentration Time Curve From Time Zero to 168 (AUC[0-168]) of TTI-621
Description: Results for this outcome measure was reported for Part 2 and Part 3 combined.
Time Frame: Part 2 and 3: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: PK -evaluable set included treated participants with adequate blood sampling to estimate at least one PK parameter. Here, "Number of participants analyzed" signifies number of evaluable participants for this outcome measure. Data for only those arms [according to dose] are reported for this outcome measure which had any evaluable participants.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter
Arm/Group | Part 2 and 3 Combined: 0.1 mg/kg | Part 2 and 3 Combined: 0.2 mg/kg | Part 2 and 3 Combined: 0.3 mg/kg | Part 2 and 3 Combined: 0.4 mg/kg | Part 2 and 3 Combined: 0.5 mg/kg
Number analyzed (Participants) | 36 | 133 | 0 | 1 | 0
Nanogram*hour per milliliter | 9330 (10300) | 20000 (10400) |  | 16100 |

12. Secondary Outcome: Part 2 and 3 Combined: Percentage of CD47 Receptor Occupancy on Peripheral Blood CD3+ Cells
Description: CD47 is a cell-surface protein expressed on multiple normal cell types and often at high levels on many malignant tumour cells. Results are reported for combined Part 2 and 3.
Time Frame: Part 2 and 3: Week 1 end of infusion (EOI)
Population: Safety population included all the participants who received at least one dose of study treatment. Here, "Number of participants analyzed" signifies number of evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of Cells
Groups:
- Part 2 and 3 Combined: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.1 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
- Part 2 and 3 Combined: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg: Participants with advanced relapsed or refractory lymphomas received TTI-621 0.2 mg/kg infusion once weekly until disease progression, unacceptable toxicity, or other reasons for treatment discontinuation occurred.
Arm/Group | Part 2 and 3 Combined: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 2 and 3 Combined: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg
Number analyzed (Participants) | 33 | 113
Percentage of Cells | 24.99 (16.54) | 31.39 (17.28)

13. Secondary Outcome: Part 2 and 3: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb)
Description: A participant was ADA (or NAb) positive if: (1) baseline titer was missing or negative and participants had >1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a > 4-fold dilution increase in titer from baseline in > 1 post-treatment sample (treatment-boosted).
Time Frame: Part 2 and 3: From pre-infusion on day 1 up to end of study treatment (maximum treatment exposure for Part 2 was 1793 days and for Part 3 was 938 days)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy
Number analyzed (Participants) | 94 | 11 | 36 | 37
Participants
  ADA Positive: Overall Incidence | 14 | 0 | 1 | 5
  NAb Positive: Overall Incidence | 1 | 0 | 0 | 0

14. Secondary Outcome: Part 2 and 3: Overall Response Rate (ORR) - Lugano Classification (Cheson 2014) and Refinement (Cheson 2016) Disease Indications and Nivolumab/Rituximab Combinations
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete remission and partial remission. Lugano classification (Cheson et al., 2014) and refinement (Cheson et al., 2016) were used for tumor response assessment for lymphomas by computed tomography (CT)-based criteria and complete metabolic response (CMR) or partial metabolic response (PMR) by positron emission tomography (PET-CT) based criteria were used for evaluation. Lymphomas evaluated by Lugano Classification include aggressive B-cell lymphoma (ABCL), Hodgkin's lymphoma (HL), Non-Hodgkin's lymphoma, indolent B-cell lymphoma (IBCL), peripheral T-cell lymphoma (PTCL), and part of T-cell lymphoma (TCL).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: Full analysis set included all participants who received at least 1 dose of study treatment. "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Aggressive B-cell Lymphoma (ABCL): Participants with ABCL who received study drug in Part 2.
- Part 2: Hodgkin Lymphoma (HL): Participants with HL who received study drug in Part 2.
- Part 2: Indolent B-cell Lymphoma (IBCL): Participants with IBCL who received study drug in Part 2.
- Part 2: Classical Hodgkin's Lymphoma (cHL): Participants with cHL who received nivolumab combination in Part 2.
- Part 2: CD20-positive Malignancies: Participants with CD20-positive malignancies who received rituximab combination in Part 2.
- Parts 2 and 3: Peripheral T-cell Lymphoma (PTCL): Participants with PTCL who received study drug in Parts 2 and 3.
- Parts 2 and 3: T-cell Lymphoma (TCL): Participants with TCL who received study drug and response assessment by Lugano Classification (Cheson 2014/2016) in Parts 2 and 3.
Arm/Group | Part 2: Aggressive B-cell Lymphoma (ABCL) | Part 2: Hodgkin Lymphoma (HL) | Part 2: Indolent B-cell Lymphoma (IBCL) | Part 2: Classical Hodgkin's Lymphoma (cHL) | Part 2: CD20-positive Malignancies | Parts 2 and 3: Peripheral T-cell Lymphoma (PTCL) | Parts 2 and 3: T-cell Lymphoma (TCL)
Number analyzed (Participants) | 5 | 13 | 5 | 11 | 40 | 21 | 11
Participants | 1 | 0 | 0 | 4 | 9 | 3 | 3

15. Secondary Outcome: Parts 2 and 3: Overall Response Rate (ORR)-Olsen 2011-Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete response and partial response. Clinical endpoints and response criteria (Olsen et al., 2011) for in CTCL (mycosis fungoides and Sezary syndrome) and TCL were used for assessment. Tumor types evaluated included Cutaneous T-cell lymphoma (CTCL) and a part of T-cell lymphoma (TCL).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Parts 2 and 3 : Cutaneous T-cell Lymphoma (CTCL): Participants with CTCL who received study drug in Parts 2 and 3.
- Parts 2 and 3: T-cell Lymphoma (TCL): Participants with TCL who received study drug and response assessment by Olsen 2011 in Parts 2 and 3.
Arm/Group | Parts 2 and 3 : Cutaneous T-cell Lymphoma (CTCL) | Parts 2 and 3: T-cell Lymphoma (TCL)
Number analyzed (Participants) | 21 | 29
Participants | 2 | 5

16. Secondary Outcome: Part 2: Overall Response Rate (ORR)-Savona 2015- Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete remission, partial remission and marrow response. International Consortium Proposal of Uniform Response Criteria for Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN) in adults (Savona et al., 2015) was used for assessment of tumors. Tumor types evaluated include Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Myelodysplastic Syndrome (MDS): Participants with MDS who received study drug in part 2.
- Part 2: Myeloproliferative Neoplasms (MPN): Participants with MPN who received study drug in part 2.
Arm/Group | Part 2: Myelodysplastic Syndrome (MDS) | Part 2: Myeloproliferative Neoplasms (MPN)
Number analyzed (Participants) | 6 | 3
Participants | 0 | 1

17. Secondary Outcome: Part 2: Overall Response Rate (ORR)- Hallek 2008- Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete response or complete remission, complete response or complete remission with incomplete marrow recovery, partial response. International Workshop on CLL update of the NCI 1996 Guidelines (Hallek et al., 2008) was used for assessment of tumors. Tumor types evaluated include chronic lymphocytic leukemia (CLL).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Chronic Lymphocytic Leukemia (CLL): Participants with CLL who received study drug in part 2.
Arm/Group | Part 2: Chronic Lymphocytic Leukemia (CLL)
Number analyzed (Participants) | 3
Participants | 0

18. Secondary Outcome: Part 2: Overall Response Rate (ORR)- Durie 2006- Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete response, stringent complete response, very good partial response, partial response. International Uniform Response Criteria for Multiple Myeloma (Durie et al., 2006). was used for assessment of tumors.Tumor types evaluated include Multiple Myeloma (MM).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Multiple Myeloma (MM): Participants with MM who received study drug in part 2.
Arm/Group | Part 2: Multiple Myeloma (MM)
Number analyzed (Participants) | 8
Participants | 0

19. Secondary Outcome: Part 2: Overall Response Rate (ORR)- Cheson 2003- Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had morphologic leukemia-free state, morphologic complete remission, morphologic complete remission with incomplete blood count recovery, partial remission. International Working Group for trials in AML (Cheson et al., 2003) was used for assessment of tumor. Tumor types evaluated include Acute Myeloid Leukemia (AML).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Acute Myeloid Leukemia (AML): Participants with AML who received study drug in part 2.
Arm/Group | Part 2: Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 20
Participants | 2

20. Secondary Outcome: Part 2: Overall Response Rate (ORR)- Bohnsack 2014- Disease Indication
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had irComplete Response, IrPartial Response. Immune-Related Response Criteria: RECIST (Bohnsack et al., 2014) was used for assessment of tumor. Tumor types evaluated included Small Cell Lung Cancer (SCLC).
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Small Cell Lung Cancer (SCLC): Participants with SCLC who received study drug in part 2.
Arm/Group | Part 2: Small Cell Lung Cancer (SCLC)
Number analyzed (Participants) | 4
Participants | 0

21. Secondary Outcome: Parts 2 and 3: Duration of Response (DoR)- Disease Indication and Nivolumab/Rituximab Combinations
Description: DoR was defined, in participants who achieved a response as time from the first date of response to the first date of recurrent or progression disease. Participants without recurrent or progression disease were censored on date of the last adequate disease assessment, date of initiation of anticancer treatment or death of death, whichever was the earliest.
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2: Aggressive B-cell Lymphoma (ABCL): Participants with ABCL who received study drug in Part 2. Response included complete remission and partial remission. Lugano Classification (Cheson et al., 2014) and refinement (Cheson et al., 2016) used for assessment.
- Part 2: Acute Myeloid Leukemia (AML): Participants with AML who received study drug in Part 2. Response included morphologic leukemia-free state, morphologic complete remission, morphologic complete remission with incomplete blood count recovery, partial remission. International Working Group for trials in AML (Cheson et al., 2003) was used for assessment.
- Part 2: Chronic Lymphocytic Leukemia (CLL): Participants with CLL who received study drug in Part 2. Response included complete response or complete remission, complete response or complete remission with incomplete marrow recovery, partial response. International Workshop on CLL update of the NCI 1996 Guidelines (Hallek et al., 2008) was used for assessment.
- Part 2: Hodgkin Lymphoma (HL): Participants with HL who received study drug in Part 2. Response included complete remission and partial remission. Lugano Classification (Cheson et al., 2014) and refinement (Cheson et al., 2016) used for assessment.
- Part 2: Indolent B-cell Lymphoma (IBCL): Participants with IBCL who received study drug in Part 2. Response included complete remission and partial remission. Lugano Classification (Cheson et al., 2014) and refinement (Cheson et al., 2016) used for assessment.
- Part 2: Myelodysplastic Syndrome (MDS): Participants with MDS who received study drug in Part 2. Response included complete remission, partial remission, marrow response. International Consortium Proposal of Uniform Response Criteria for Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN) in Adults (Savona et al., 2015) was used for assessment.
- Part 2: Multiple Myeloma (MM): Participants with MM who received study drug in Part 2. Response included complete response, stringent complete response, very good partial response, partial response. International Uniform Response Criteria for Multiple Myeloma (Durie et al., 2006) was used for assessment.
- Part 2: Myeloproliferative Neoplasms (MPN): Participants with MPN who received study drug in Part 2. Response included complete remission, partial remission, marrow response. International Consortium Proposal of Uniform Response Criteria for Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN) in Adults (Savona et al., 2015) was used for assessment.
- Part 3: Peripheral T-cell Lymphoma (PTCL): Participants with PTCL who received study drug in Part 3. Response included complete remission and partial remission. Lugano Classification (Cheson et al., 2014) and refinement (Cheson et al., 2016) used for assessment.
- Part 2: Small Cell Lung Cancer (SCLC): Participants with SCLC who received study drug in part 2. Response included irComplete Response, irPartial Response. Immune-Related Response Criteria: irRECIST (Bohnsack et al., 2014) was used for assessment.
- Parts 2 and 3: Cutaneous T-cell Lymphoma (CTCL): Participants with CTCL who received study drug in Parts 2 and 3. Response included complete response, partial response. Clinical endpoints and response criteria (Olsen et al., 2011) were used in CTCL (mycosis fungoides and Sezary syndrome).
- Parts 2 and 3: T-cell Lymphoma (TCL): Participants with TCL who received study drug in Parts 2 and 3. Response included complete remission and partial remission. Response criteria included both Lugano Classification (Cheson 2014/ refinement 2016) and Olsen 2011 used for assessment.
Arm/Group | Part 2: Aggressive B-cell Lymphoma (ABCL) | Part 2: Acute Myeloid Leukemia (AML) | Part 2: Chronic Lymphocytic Leukemia (CLL) | Part 2: Hodgkin Lymphoma (HL) | Part 2: Indolent B-cell Lymphoma (IBCL) | Part 2: Myelodysplastic Syndrome (MDS) | Part 2: Multiple Myeloma (MM) | Part 2: Myeloproliferative Neoplasms (MPN) | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 3: Peripheral T-cell Lymphoma (PTCL) | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Part 2: Small Cell Lung Cancer (SCLC) | Parts 2 and 3: Cutaneous T-cell Lymphoma (CTCL) | Parts 2 and 3: T-cell Lymphoma (TCL)
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 9 | 0 | 2 | 8
Months | NA [NA to NA] — Median and 95% CI could not be estimated due to less number of participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to less number of participants with events. |  |  |  |  |  | 8.3 [NA to NA] — 95% CI could not be estimated due to less number of participants with events. | 9.2 [NA to NA] — 95% CI could not be estimated due to less number of participants with events. | 12.0 [NA to NA] — 95% CI could not be estimated due to less number of participants with events. | 3.1 [1.9 to 21.3] |  | 1.9 [1.8 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 8.3 [1.0 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events.

22. Secondary Outcome: Parts 2 and 3: Progression Free Survival (PFS)
Description: PFS was defined as the number of weeks from the date of the first dose of study drug to the earliest of documented recurrent or progressive disease or death due to any cause without prior progression. The progression or censoring date was determined based on described conventions (Food and Drug Administration, 2007). Kaplan-Meier method was used.
Time Frame: From first dose of study till the progressive disease/ death or withdrawal (maximum observation 6 years 10 months)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2: Chronic Lymphocytic Leukemia (CLL): Participants with CLL who received study drug in Part 2. Response included complete response or complete remission, complete response or complete remission with incomplete marrow recovery, partial response. International Workshop on CLL update of the NCI 1996 Guidelines Chronic lymphocytic leukemia (CLL) Participants with (CLL) NOTE: An Arm/Group Description is shorter than the Arm/Group Title. Response included complete response or complete remission, complete response or complete remission with incomplete marrow recovery, partial response. International Workshop on CLL update of the NCI 1996 Guidelines (Hallek et al., 2008) was used for assessment.
Arm/Group | Part 2: Aggressive B-cell Lymphoma (ABCL) | Part 2: Acute Myeloid Leukemia (AML) | Part 2: Chronic Lymphocytic Leukemia (CLL) | Part 2: Hodgkin Lymphoma (HL) | Part 2: Indolent B-cell Lymphoma (IBCL) | Part 2: Myelodysplastic Syndrome (MDS) | Part 2: Multiple Myeloma (MM) | Part 2: Myeloproliferative Neoplasms (MPN) | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 3: Peripheral T-cell Lymphoma (PTCL) | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Part 2: Small Cell Lung Cancer (SCLC) | Parts 2 and 3: Cutaneous T-cell Lymphoma (CTCL) | Parts 2 and 3: T-cell Lymphoma (TCL)
Number analyzed (Participants) | 3 | 17 | 2 | 9 | 3 | 5 | 8 | 2 | 5 | 14 | 37 | 0 | 9 | 22
Months | 1.6 [0.7 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 0.8 [0.7 to 1.0] | 1.4 [0.8 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 3.1 [1.0 to 4.4] | 1.4 [0.7 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 0.8 [0.7 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 1.1 [0.7 to 1.3] | 11.0 [5.6 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 3.5 [0.7 to NA] — Upper limit of 95% CI could not be estimated due to less number of participants with events. | 1.7 [1.5 to 3.1] | 1.7 [1.5 to 2.3] |  | 5.4 [1.9 to 10.8] | 2.6 [1.6 to 15.8]

23. Secondary Outcome: Part 4: Maximum Plasma Concentration (Cmax) of TTI-621
Time Frame: Part 4: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: The Pharmacokinetic (PK)-evaluable Set consists of treated participants with adequate blood sampling to estimate at least one pharmacokinetic PK parameter. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 10 | 1
Nanogram per milliliter | 4040 (110) | 6190 (1100) | 10000 (4400) | 15400 (2470) | 23600 (4530) | 18800

24. Secondary Outcome: Part 4: Area Under the Plasma Concentration Time Curve From Time Zero to 168 (AUC[0-168]) of TTI-621
Time Frame: Part 4: Pre-dose, end of infusion (EOI), 2, 4, 24, 72, 168 hours post dose on Week 1
Population: PK -evaluable set included treated participants with adequate blood sampling to estimate at least one PK parameter. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 8 | 0
Nanogram*hour per milliliter | 88800 (12300) | 116000 (38800) | 212000 (85700) | 383000 (49600) | 638000 (120000) |

25. Secondary Outcome: Part 4: Percentage of CD47 Receptor Occupancy on Peripheral Blood CD3+ Cells
Description: CD47 is a cell-surface protein expressed on multiple normal cell types and often at high levels on many malignant tumor cells.
Time Frame: Part 4: Week 1 end of infusion (EOI)
Population: Safety population included all the participants who received at least one dose of study treatment. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 3
Percentage of cells | 62.25 (12.65) | 65.49 (24.80) | 37.17 (32.93) | 57.09 (23.72) | 65.00 (5.97) | 49.51 (10.83)

26. Secondary Outcome: Part 4: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb)
Description: A participant was ADA (or NAb) positive if: (1) baseline titer is missing or negative and participants had >1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a > [4-fold dilution increase] in titer from baseline in > 1 post-treatment sample (treatment-boosted).
Time Frame: Part 4: From pre-infusion on day 1 up to end of study treatment (maximum treatment exposure for Part 4 was 667 days)
Population: Immunogenicity analysis population includes all treated participants with at least one (ADA) Anti-Drug Antibody sample (pre-dose or post-treatment) analyzed. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 11 | 4
Participants
  ADA Positive: Overall Incidence | 0 | 0 | 0 | 0 | 0 | 0
  NAb Positive: Overall Incidence | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Part 4: Overall Response Rate (ORR)
Description: ORR is presented in this outcome measure as number of responders. Responders were those who had complete response, partial response. Lymphomas evaluated include Non-Hodgkin's Lymphoma. Clinical endpoints and response criteria in mycosis fungoides and Sezary syndrome (Olsen et al., 2011).
Time Frame: From first dose of study till the progressive disease/death or withdrawal (maximum observation 6 years 10 months)
Population: Analysis population included all the participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 4
Participants | 0 | 0 | 1 | 1 | 2 | 0

28. Secondary Outcome: Part 4: Duration of Response (DoR)
Description: as for outcome 21
Time Frame: From first dose of study till the progressive disease/death or withdrawal (maximum observation 6 years 10 months)
Population: Analysis population included all the participants who received at least one dose of study treatment. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 2 | 0
Months |  |  | NA [NA to NA] — Median and 95% CI could not be estimated due to less number of participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to less number of participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to less number of participants with events. |

29. Secondary Outcome: Part 4: Overall Response Rate (ORR) in Cutaneous T-Cell Lymphoma (CTCL) Both Fungoides and Sezary Syndrome
Description: ORR is presented in this outcome measure as number of responders.
Time Frame: From first dose of study till the progressive disease/death or withdrawal (maximum observation 6 years 10 months)
Population: Data for this outcome measure is not available as analysis was not performed because: 1) due to futility and heterogenicity of respective data of the parameters of organ system (i.e., skin, blood, lymph node, and viscera; 2) the Olsen 2011 criteria already defined the "Global Response Score" to determine the Global Response (GR) consisting of the 4 components which (GR) was more important assessment affecting overall prognosis.
Groups:
- Part 4: CTCL: Participants with CTCL who received study drug in part 4.
Arm/Group | Part 4: CTCL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 30 days after last dose (maximum treatment exposure for: Part 1 was 414 days, Part 2 was 1793 days, Part 3 was 938 days, and Part 4 was 667 days)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis population included all the participants who received at least one dose of study treatment.
Arm/Group | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/7 | 1/5 | 52/107 | 0/11 | 27/40 | 16/42 | 0/3 | 0/3 | 2/6 | 0/3 | 5/12 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/7 | 2/5 | 43/107 | 2/11 | 13/40 | 15/42 | 1/3 | 1/3 | 2/6 | 0/3 | 3/12 | 3/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 7/7 | 5/5 | 100/107 | 11/11 | 34/40 | 36/42 | 3/3 | 2/3 | 6/6 | 3/3 | 12/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg (N=3) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg (N=3) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg (N=7) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg (N=5) | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy (N=107) | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination (N=11) | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination (N=40) | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy (N=42) | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg (N=6) | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg (N=12) | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg (N=4)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Erythroid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Graft Versus Host Disease (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophagocytic Lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza A Virus Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intramedullary Rod Insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.05 mg/kg (N=3) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.1 mg/kg (N=3) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.2 mg/kg (N=7) | Part 1: Ontorpacept (PF-07901800/TTI-621) 0.3 mg/kg (N=5) | Part 2: Ontorpacept (PF-07901800/TTI-621) Monotherapy (N=107) | Part 2: Ontorpacept (PF-07901800/TTI-621)+ Nivolumab Combination (N=11) | Part 2: Ontorpacept (PF-07901800/TTI-621) + Rituximab Combination (N=40) | Part 3: Ontorpacept (PF-07901800/TTI-621) Monotherapy (N=42) | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.5 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 0.7 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.0 mg/kg (N=6) | Part 4: Ontorpacept (PF-07901800/TTI-621) 1.4 mg/kg (N=3) | Part 4: Ontorpacept (PF-07901800/TTI-621) 2.0 mg/kg (N=12) | Part 4: Ontorpacept (PF-07901800/TTI-621) Q2W / 2.0 mg/kg (N=4)
Fatigue (General disorders) | 1 | 2 | 4 | 2 | 39 | 0 | 18 | 13 | 1 | 0 | 1 | 0 | 4 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 28 | 5 | 5 | 16 | 0 | 0 | 2 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 23 | 3 | 10 | 10 | 1 | 1 | 2 | 0 | 2 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 9 | 2 | 5 | 4 | 0 | 0 | 2 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 2 | 4 | 4 | 44 | 5 | 17 | 14 | 1 | 2 | 4 | 2 | 5 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 11 | 0 | 3 | 5 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 28 | 3 | 8 | 6 | 0 | 1 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 3 | 23 | 2 | 8 | 5 | 0 | 1 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 20 | 2 | 7 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 11 | 3 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 31 | 4 | 10 | 8 | 0 | 0 | 0 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 23 | 3 | 6 | 6 | 0 | 1 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 7 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 12 | 1 | 9 | 5 | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 12 | 1 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 8 | 6 | 0 | 5 | 0 | 0 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 6 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 20 | 3 | 7 | 10 | 0 | 0 | 1 | 1 | 8 | 1
Neutrophil Count Decreased (Investigations) | 0 | 0 | 1 | 0 | 8 | 0 | 4 | 2 | 0 | 0 | 0 | 1 | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 20 | 4 | 4 | 5 | 0 | 0 | 2 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 16 | 0 | 3 | 6 | 0 | 0 | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 17 | 1 | 3 | 9 | 1 | 0 | 1 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 14 | 0 | 8 | 6 | 1 | 0 | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 15 | 0 | 5 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 15 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 11 | 1 | 4 | 8 | 1 | 2 | 2 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 5 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 14 | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 7 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 12 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 10 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02663518/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT02663518/SAP_001.pdf